CLINICAL TRIAL: NCT04818840
Title: A Prospective Multi-Centre Study in Patients Undergoing Total Knee Replacement With JOURNEY II CR Total Knee System
Brief Title: Evaluate the Performance of JOURNEY II CR in TKA Populations
Acronym: JIICRTKA
Status: Terminated | Type: Observational
Why Stopped: It was terminated by sponsor for updated evidence needs
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Journey II CR.2020.11
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-08

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Osteoarthritis; Total knee arthroplasty (TKA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Resurfaced/non patella: Undergoing Total Knee Replacement with JOURNEY II CR Total Knee System
  Interventions: Device: Resurfaced Patella
- un-resurfaced patella: Undergoing Total Knee Replacement with JOURNEY II CR Total Knee System
  Interventions: Procedure: Un-resurfaced Patella

INTERVENTIONS:
Device: Resurfaced Patella — JOURNEY II CR Total Knee System was used for Total Knee replacement
  Groups: Resurfaced/non patella
Procedure: Un-resurfaced Patella — JOURNEY II CR Total Knee System was used for Total Knee replacement
  Groups: un-resurfaced patella

SUMMARY:
Background:

The JOURNEY II CR Total Knee System consists of femoral component made from oxidized zirconium (OXINIUM)

Purpose:

Post-market evidence generation for JOURNEY II CR Total Knee System

Objectives:

Evaluate the performance of JOURNEY II CR TKA in APAC populations Evaluate the impact of patella resurfacing on the outcomes of JOURNEY II CR TKA

Research participants / locations:

A total of up to 480 knees' information will be collected in up to 15 sites in India, China mainland, Hong Kong, Singapore, Thailand and Japan There will be up to 240 knees for resurfaced patella group and up to 240 knees for un-resurfaced patella group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with degenerative osteoarthritis.
* Subject is planning to have TKA using JOURNEY II CR.
* Subject is able and willing to provide voluntary consent to study participation.
* Subject is 18-80 years old (inclusive) * (* For Japan, the minimum inclusion age is 20 years old.)

Exclusion Criteria:

* Subjects with rheumatoid arthritis/inflammatory arthritis, posttraumatic arthritis.
* Previous surgeries including HTO, UKA or TKA on the subject knee.
* Subject is pregnant or breast feeding or those at a child-bearing age planning to become pregnant during the follow up.
* Subject does not meet the indication or is contraindicated for JOURNEY II CR's IFU.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of up to 480 knees' information will be collected in up to 15 sites in India, China mainland, Hong Kong, Singapore, Thailand and Japan There will be up to 240 knees for resurfaced patella group and up to 240 knees for un-resurfaced patella group.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Yang, Study Director — Smith & Nephew, Inc.
Locations (8):
- China (2):
  - Peking University Third Hospital, Beijing
  - Prince of Wales Hospital, Hong Kong
- India (2):
  - Aster RV Hospital, Bangalore, Bengaluru, Karnataka
  - Arcus Hospital, Pune, Maharashtra
- Japan (2):
  - Toho University Omori Medical Center, Tokyo
  - Tokyo Women's Medical University, Tokyo
- Singapore General Hospital, Singapore, Singapore
- Chulalongkorn Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 62 participants in total enrolled into the study across 5 study sites. The 60 participants that received the study device were included in the analysis. Two participants were excluded before assignment to groups because they did not receive the study device.
Period: Overall Study
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Started | 44 | 16
Completed | 0 | 0
Not Completed | 44 | 16
Not completed — Lost to Follow-up | 0 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Site Terminated by Sponsor | 0 | 3
Not completed — Study Terminated by Sponsor | 43 | 7
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella | Total
Number analyzed (Participants) | 44 | 16 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 34 | 12 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.0) | 68.0 (6.8) | 69.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 11 | 45
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 44 | 16 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 0 | 3 | 3
  Japan | 43 | 0 | 43
  China | 0 | 10 | 10
  Hong Kong | 1 | 3 | 4
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 155.7 (7.6) | 157.6 (9.5) | 156.2 (8.1)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 67.5 (15.5) | 67.4 (8.7) | 67.5 (13.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.6) | 27.2 (2.8) | 27.5 (4.2)
Operative Diagnosis [Count of Participants; unit: Participants]
  Osteoarthritis | 43 | 16 | 59
  Avascular necrosis | 1 | 0 | 1
  Functional deformity | 0 | 0 | 0
  Fractures that were unmanageable using other techniques | 0 | 0 | 0
  Missing | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score (OKS) at 2 Years
Description: The Oxford Knee Score (OKS) is a Patient Reported Outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty (TKA). The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Time Frame: 2 years
Population: Data not collected for outcome because no participant reached the 2 year time frame due to early termination of the study. While the general study duration does cover 2 years, there were multiple sites. No participant at any site reached the 2 year time point because the study was terminated before any of the data was collected for this visit.
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The Forgotten Joint Score (FJS) comprises measures for the assessment of joint-specific patient reported outcomes. This questionnaire focuses on the study participant's awareness of the partially or fully replaced knee joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. Participants are asked to rate their awareness of their knee arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living (i.e., a higher score is a better outcome).
Time Frame: 6 months, 1 year, 2 years, 3 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. Data not collected for all time points due to early termination of the study. While the general study duration does cover 2 years, there were multiple sites. No participant at any site reached the 2 year time point because the study was terminated before any of the data was collected for any visit on or after the 2 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 27 | 9
score on a scale
  6 months | 40.8 (22.2) | 72.2 (30.4)
  1 year: number analyzed (Participants) | 22 | 4
  1 year | 49.0 (28.6) | 89.6 (20.8)
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Oxford Knee Score (OKS)
Description: The Oxford Knee Score (OKS) is a Patient Reported Outcome (PRO) questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty (TKA). The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Overall scores range from 0 to 48, where a score of 0 is the worst possible outcome and a score of 48 is the best possible outcome.
Time Frame: Pre-Operative, 6 months, 1 year, 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 42 | 16
score on a scale
  Pre-Operative | 21.0 (9.1) | 22.9 (7.8)
  6 months: number analyzed (Participants) | 29 | 9
  6 months | 35.2 (8.2) | 37.3 (10.0)
  1 year: number analyzed (Participants) | 21 | 4
  1 year | 38.0 (7.6) | 44.5 (4.4)
  3 years: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Knee Society Score (KSS): "Objective" Knee Score
Description: The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales: The "Objective" Knee Score sub-scale is assessed by the surgeon, focusing on clinical measures such as pain, range of motion, and stability. The score is 7 items on a scale of 0 to 100 where a higher score indicates a better outcome.
Time Frame: Pre-Operative, 6 months, 1 year, 2 years, 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 42 | 5
score on a scale
  Pre-Operative | 23.6 (20.6) | 28.6 (12.3)
  6 months: number analyzed (Participants) | 26 | 3
  6 months | 70.0 (7.4) | 68.7 (8.0)
  1 year: number analyzed (Participants) | 21 | 0
  1 year | 72.5 (7.3) |
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Knee Society Score (KSS): Patient Satisfaction Score
Description: The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales. The Patient Satisfaction sub-scale score evaluates the participant's satisfaction with their knee function and pain relief. The score is five items on a scale of 0 to 40 where a higher score indicates a better outcome.
Time Frame: Pre-Operative, 6 months, 1 year, 2 years, 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 42 | 16
score on a scale
  Pre-Operative | 11.7 (7.5) | 11.4 (9.2)
  6 months: number analyzed (Participants) | 27 | 9
  6 months | 22.7 (8.1) | 28.9 (4.9)
  1 year: number analyzed (Participants) | 22 | 4
  1 year | 28.0 (8.5) | 31.0 (6.6)
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Knee Society Score (KSS): Patient Expectation Score
Description: The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales. The Patient Expectation sub-scale score assesses the participant's expectations regarding their knee function and outcomes. The score is three items on a scale of 3 to 15 where a higher score indicates a better outcome.
Time Frame: Pre-Operative, 6 months, 1 year, 2 years, 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 42 | 16
score on a scale
  Pre-Operative | 13.8 (1.5) | 14.4 (2.0)
  6 months: number analyzed (Participants) | 27 | 9
  6 months | 9.0 (3.0) | 11.0 (3.1)
  1 year: number analyzed (Participants) | 22 | 4
  1 year | 9.7 (2.9) | 10.3 (2.5)
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Knee Society Score (KSS): Functional Knee Score
Description: The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales. The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities to evaluate the participant's ability to perform daily activities and their overall functional capabilities. The score is 19 items on a scale of 0 to 100 where a higher score indicates a better outcome.
Time Frame: Pre-Operative, 6 months, 1 year, 2 years, 3 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 17 | 6
score on a scale
  Pre-Operative | 47.8 (20.0) | 47.2 (15.1)
  6 months: number analyzed (Participants) | 7 | 5
  6 months | 80.4 (7.2) | 86.2 (14.5)
  1 year: number analyzed (Participants) | 6 | 4
  1 year | 83.8 (21.0) | 89.8 (11.5)
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Expectation
Description: Patient expectation measured by asking participants to select "ONE activity that matters to you most and you expect to participate after the surgery?" Responses were categorized as:
  1. Regularly participate in impact sports (e.g., jogging, tennis, skiing, acrobatics, ballet, heavy labor, backpacking, basketball, mountain climbing or badminton with running & jumping)
  2. Sometime participate in impact sports
  3. Regularly participate in very active events (e.g., bowling, golf, table tennis, badminton without running & jumping or fitness walking)
  4. Regularly participate in active events (e.g., bicycling or square dancing)
  5. Regularly participate in moderate activities (e.g., swimming & unlimited housework, shopping or Tai Chi)
  6. Sometimes participate in moderate activities
  7. Regularly participate in mild activities (e.g., walking, limited housework, & limited shopping)
  8. Sometimes participate in mild activities
  9. Restricted to minimal activities of daily living
  10. Missing
Time Frame: Pre-Operative
Population: Participants that received the study device with data collected for the outcome and time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 44 | 16
Participants
  Regularly participate in impact sports | 5 | 1
  Sometime participate in impact sports | 0 | 1
  Regularly participate in very active events | 4 | 0
  Regularly participate in active events | 0 | 4
  Regularly participate in moderate activities | 14 | 5
  Sometimes participate in moderate activities | 2 | 0
  Regularly participate in mild activities | 8 | 5
  Sometimes participate in mild activities | 1 | 0
  Restricted to minimal activities of daily living | 1 | 0
  Missing | 9 | 0

9. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction is measured by a corresponding question based on their expectation asking, "How satisfied are you with the surgery meeting your expectation?" Responses were categorized as:
  * Very Satisfied
  * Satisfied
  * Neutral
  * Dissatisfied
  * Very Dissatisfied
  * Missing
Time Frame: 6 months, 1 year, 2 years, 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 34 | 9
Participants
  6 months: Very Satisfied | 4 | 3
  6 months: Satisfied | 12 | 3
  6 months: Neutral | 5 | 3
  6 months: Dissatisfied | 1 | 0
  6 months: Very Dissatisfied | 0 | 0
  6 months: Missing | 12 | 0
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Very Satisfied | 5 | 1
  1 year: Satisfied | 10 | 3
  1 year: Neutral | 4 | 0
  1 year: Dissatisfied | 1 | 0
  1 year: Very Dissatisfied | 1 | 0
  1 year: Missing | 6 | 0
  2 years: number analyzed (Participants) | 0 | 0
  3 years: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Radiographic Assessment: Presence of Radiographic Findings
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the number of participants with the presence of radiographic findings categorized as:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 10
  Immediate Post-Op to 6 weeks: No | 43 | 6
  Immediate Post-Op to 6 weeks: Missing | 0 | 0
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 1 | 6
  6 months: No | 33 | 3
  6 months: Missing | 3 | 0
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 3
  1 year: No | 25 | 1
  1 year: Missing | 2 | 0
  2 years: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Radiographic Assessment: Aseptic Loosening
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of aseptic loosening as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from a site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for Aseptic Loosening radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Radiographic Assessment: Septic Loosening
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of septic loosening as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from a site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Septic Loosening radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Radiographic Assessment: Bone Fracture
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of bone fracture as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from one site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Bone Fracture radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Radiographic Assessment: Cement Fracture
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of cement fracture as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from one site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Cement Fracture radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Radiographic Assessment: Osteolysis
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of osteolysis as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from one site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Osteolysis radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Radiographic Assessment: Subsidence
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of subsidence as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from one site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Subsidence radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Radiographic Assessment: Implant Migration
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of implant migration as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from a site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Implant Migration radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Radiographic Assessment: Stress Shielding
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of stress shielding as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from a site indicated radiographic findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Stress Shielding radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 1 | 0
  6 months: No | 0 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Radiographic Assessment: Implant-Cement Debonding
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to identify the radiographic finding type by the presence of implant-cement debonding as one of the following:
  * Yes
  * No
  * Missing
Time Frame: Immediate Post-op to 6 weeks, 6 months, 1 year, 2 years
Population: Participants that received the study device with data collected for the outcome and time frame indicated. While general study duration covers 2 years, there were multiple sites with no participant reaching the 2 year visit for data collection due to study termination. Responses from a site indicated findings for participants in the un-resurfaced patella group (i.e., "Yes" to presence of radiographic findings), but 'No' indicated for the Implant-Cement Debonding radiographic finding option.
Measure: Count of Participants; unit: Participants
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 43 | 16
Participants
  Immediate Post-Op to 6 weeks: Yes | 0 | 0
  Immediate Post-Op to 6 weeks: No | 0 | 10
  Immediate Post-Op to 6 weeks: Missing | 43 | 6
  6 months: number analyzed (Participants) | 37 | 9
  6 months: Yes | 0 | 0
  6 months: No | 1 | 6
  6 months: Missing | 36 | 3
  1 year: number analyzed (Participants) | 27 | 4
  1 year: Yes | 0 | 0
  1 year: No | 0 | 3
  1 year: Missing | 27 | 1
  2 years: number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Radiographic Assessment: Mechanical Axis Alignment of the Knee Joint
Description: Standard radiographic evaluation on antero-posterior (A/P) and lateral views performed to determine mechanical axis alignment of the knee joint in degrees measured through the centre of the hip (centre of the spherical femoral head), centre of the knee (centre of the tibial plateau) and centre of the ankle (centre of the talus).
Time Frame: Pre-Operative, 6 months, 1 year, 2 years
Population: While general study duration does cover 2 years, there were multiple sites. No participant at any site reached the 2 year time point because the study was terminated before any of the data was collected for any visit on or after the 2 year visit. Additionally, 0 participants were analyzed at 1 year for mechanical axis alignment because data was not provided by the third party central imaging lab due to contract suspension and later study termination, so data after 6 months cannot be reported.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
Number analyzed (Participants) | 44 | 16
degrees
  Pre-Operative | 7.1 (5.1) | 9.6 (6.4)
  6 months: number analyzed (Participants) | 34 | 9
  6 months | 1.5 (1.7) | 1.5 (1.4)
  1 year: number analyzed (Participants) | 0 | 0
  2 years: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from surgery to study termination, approximately 1 year.
Arm/Group | Resurfaced/Non Patella | Un-resurfaced Patella
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/44 | 2/16
Other Adverse Events (participants affected / at risk) | 20/44 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resurfaced/Non Patella (N=44) | Un-resurfaced Patella (N=16)
OSTEOARTHRITIS IN THE CARPOMETACARPAL JOINT OF THE RIGHT THUMB (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
ACUTE GALLBLADDER INFLAMMATION (Hepatobiliary disorders) | 1 | 0 — Not related to device or procedure
LOCALIZED PROSTATE CANCER (Reproductive system and breast disorders) | 1 | 0 — Not related to device or procedure
STERNUM FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
LEFT BREAST CANCER (Reproductive system and breast disorders) | 1 | 0 — Not related to device or procedure
LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
PAIN AND SWELLING DYSFUNCTION AFTER RIGHT KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to device but related to procedure
PAIN AFTER RIGHT KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to device or procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resurfaced/Non Patella (N=44) | Un-resurfaced Patella (N=16)
FEVER (General disorders) | 3 | 0 — Not related to device or procedure
UTERINE MYOMA (Reproductive system and breast disorders) | 1 | 0 — Not related to device or procedure
ILIOTIBIAL BAND SYNDROME OF RIGHT LEG (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
NUMBNESS IN RIGHT TOES (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
RIGHT OTITIS MEDIA WITH EFFUSION (Ear and labyrinth disorders) | 1 | 0 — Not related to device or procedure
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 — Not related to device or procedure
DIZZINESS (General disorders) | 1 | 0 — Not related to device or procedure
LEFT COXODYNIA (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
PRIMARY HAND ARTHROPATHY OF RIGHT HAND (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
PERIPHERAL NEUROPATHY (Nervous system disorders) | 1 | 0 — Not related to device or procedure
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 | 0 — Not related to device or procedure
LEFT LUMBALGIA (General disorders) | 1 | 0 — Not related to device or procedure
TRANSIENT LOSS OF CONSCIOUSNESS (General disorders) | 1 | 0 — Not related to device or procedure
SEBORRHEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 — Not related to device or procedure
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
UPPER AND LOWER EXTREMITY ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 — Not related to device or procedure
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 — Not related to device or procedure
CYSTITIS (Renal and urinary disorders) | 1 | 0 — Not related to device or procedure
RIGHT ANKLE SPRAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
REFLUX ESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 — Not related to device or procedure
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 — Not related to device or procedure
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 | 0 — Not related to device or procedure
BOTH LOWER EXTREMITY ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 — Not related to device or procedure
TINNITUS (Ear and labyrinth disorders) | 1 | 0 — Not related to device or procedure
LEFT LOWER LEG CRAMPS IN THE CALVES (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to device or procedure
MALAISE (Psychiatric disorders) | 1 | 0 — Not related to device or procedure
SCIATICA (Musculoskeletal and connective tissue disorders) | 2 | 0 — Not related to device or procedure
GASTRALGIA (Gastrointestinal disorders) | 1 | 0 — Not related to device or procedure
DIZZINESS (General disorders) | 0 | 1 — Not related to device or procedure
TREMORS (Nervous system disorders) | 0 | 1 — Not related to device or procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04818840/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT04818840/SAP_001.pdf